CLINICAL TRIAL: NCT06929858
Title: Effect of Cognitive-Behavioral Strategies on Self-Efficacy, Sense of Coherence, and Psychological Ownership Among Nurses Caring for Children With Autism Spectrum Disorder
Brief Title: Effect of Cognitive-Behavioral Strategies on Nurses Caring for Children With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCBR-375/2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-12

CONDITIONS: Nurses Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBS Intervention group (Experimental): Interventional study gropu receives the cognitive-behavioral strategies training
  Interventions: Other: cognitive-behavioral strategies training
- Control (No Intervention): Continues with usual practice

INTERVENTIONS:
Other: cognitive-behavioral strategies training — A structured training program focused on cognitive-behavioral strategies tailored to the challenges of caring for children with ASD. Examples include:
  Techniques to manage stress (e.g., relaxation exercises). Cognitive reframing to address negative thoughts. Coping skills to enhance resilience in a demanding work environment.
  Arms: CBS Intervention group

SUMMARY:
The purpose of this study is to determine if a structured training program in cognitive-behavioral strategies can improve:

Self-efficacy: The belief in one's ability to succeed in specific tasks or situations.

Sense of coherence: A perception of life as comprehensible, manageable, and meaningful.

Psychological ownership: A sense of possession or attachment to one's job or role.

These outcomes are critical for nurses working with children with ASD, as their role involves unique emotional and professional challenges. The study will use a rigorous scientific approach to assess the effectiveness of the intervention.

ELIGIBILITY:
Registered nurses who provide direct care to children with ASD in settings such as hospitals, clinics, or specialized care centers.

Inclusion Criteria:

* At least 6 months of experience caring for children with ASD.
* Currently employed in a direct caregiving role for these children.

Exclusion Criteria:

* Nurses with prior formal training in cognitive-behavioral therapy.
* Nurses planning to leave their position during the study period.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy | 2 months
  Tool: Nursing Self-Efficacy Scale, Total scores range from 10 to 40, with higher scores indicating greater self-efficacy.

SECONDARY OUTCOMES:
Sense of Coherence | 2 months
  Tool: Sense of Coherence Scale, Total scores range from 13 to 91, with higher scores indicating a stronger sense of coherence.

REFERENCES:
- [Derived] Zoromba MA, Alenezi A, El-Monshed AH, Loutfy A, Ali AM, Alkubati SA, El-Gazar HE. Effect of Cognitive-Behavioural Strategies on Self-Efficacy, Sense of Coherence and Psychological Ownership Among Nurses Caring for Children With Autism Spectrum Disorder: A Randomised Control Trial. J Psychiatr Ment Health Nurs. 2026 Feb;33(1):97-108. doi: 10.1111/jpm.70066. Epub 2025 Nov 24. PMID 41277762